CLINICAL TRIAL: NCT07253350
Title: Effectiveness of Endorotor PED® System Versus Conventional Endoscopic Techniques for the Management of Walled-off Pancreatic Necrosis in Acute Necrotizing Pancreatitis: Randomized Single-blinded Controlled Superiority Trial and Cost-utility Analysis
Acronym: ROTONEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP230816; ID-RCB (Other: 2024-A01139-38)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Necrotizing Pancreatitis
Keywords: endoscopic necrosectomy; necrotic pancreatic collection
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endorotor Group (Experimental): DEN will be performed with Endorotor 3.2 or ENDOROTOR PED® system depending on the position of cystoenterostomy.
  Interventions: Device: Endorotor Group
- Conventional group (Active Comparator): DEN is performed conventionally with abundant lavage and mechanical debridement using a non-dedicated material (diathermic loop, polypectomy or Dormia basket) to catch pieces of necrosis
  Interventions: Other: Conventional group

INTERVENTIONS:
Device: Endorotor Group — DEN will be performed with Endorotor 3.2 or ENDOROTOR PED® system depending on the position of cystoenterostomy. Endorotor 3.2 is slimmer and enters WON more easily when the transgastric access is located in the upper portion of the stomach). If needed: lavage, aspiration and conventional mechanical debridement could be used in addition during an ENDOROTOR-based DEN session.
  Arms: Endorotor Group
Other: Conventional group — DEN is performed conventionally with abundant lavage and mechanical debridement using a non-dedicated material (diathermic loop, polypectomy or Dormia basket) to catch pieces of necrosis
  Arms: Conventional group

SUMMARY:
This is a national single-blinded prospective multicenter randomized (1:1) controlled trial, with two parallel arms, using a PROBE methodology, including patients with complicated acute necrotizing pancreatitis who require DEN of WON collection after endoscopic drainage. We will compare 2 groups: conventional DEN and DEN with Endorotor®. The study will be offered to all consecutive patients fulfilling the eligibility criteria after endoscopic drainage for WON. Since the time between drainage and the first necrosectomy session is usually at least 48 hours a period of at least 24h will be allowed for the patient to consider options to participate or not. Information and collection of informed consent will be done by an investigating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18years
* ASA<5
* CT scan less than 7 days old
* Hospitalized for acute necrotizing pancreatitis, whatever the cause, and who have undergone drainage of pancreatic collections for the following indications according to the revised Atlanta criteria (infection, organ compression, persistent organ failure)
* Have need for at least one DEN session despite endoscopic drainage (persistence of clinical symptoms or sepsis >48h after drainage with collection still visible)

Exclusion Criteria:

* No endoscopic drainage in place for the management of WON
* Have already had a DEN session (endoscopic or else) before screening for inclusion
* Life-expectancy < 1year (advanced cancer, etc)
* Known haemostasis disorder (chronic thrombocytopenia, haemophilia, etc.)
* Pregnant or breastfeeding woman
* Subject deprived of freedom, subject under a legal protective measure
* Non-affiliation to a social security regimen or CMU
* Patient or person of confidence (if present at the time of inclusion) opposing the patient's participation in research
* Subject already involved in another interventional clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
evaluate the effectiveness of the Endorotor PED® device versus conventional technique for the endoscopic management of symptomatic walled-off necrosis during necrotizing acute pancreatitis. | 5 month
  The effectiveness of the operative approach (Endorotor 3.2/PED® or conventional technique) will be assessed by the period in days between the first DEN session and the confirmed complete necrosis resolution.

SECONDARY OUTCOMES:
number of death | 10 month
number of new-onset multiple organ failure | 10 month
number of visceral perforation | 10 month
number of arterial perforation | 10 month
number of pancreatic-cutaneous fistulas | 10 month
number of sepsis | 10 month
number of abscess | 4 month
number of Bleeding of any severity | 4 month
number of Need for surgery (video-assisted retroperitoneal debridement or open surgery) | 4 month
number of Need for "multigate" strategy with the installation of a percutaneous drain | 4 month
time to total recovery of acute pancreatitis | 16 month
Total time of all DEN sessions in minutes | 4 month
Total number of DEN sessions | 4 month
Number of days of antibiotic treatment | 4 month
operative difficulty of DEN assessed by endoscopists | 4 month
  A Likert score will be used to assess the ease of use to maneuver device by endoscopist, from 0 (most difficult surgery imaginable) to 10 (easiest).
number of issues with Endorotor PED® device | 4 month
  Failure types and number of occurrences
Number of days of hospitalization: In intensive care unit | 16 month
Number of days of hospitalization: In conventional unit | 16 month
Number of days of hospitalization in rehabilitation unit | 16 month
quality of life of patients during and after hospitalization | 16 month
  EQ-5D-5L score at the end of hospitalization and during follow-up's visits
Total hospital costs in acute care per patient Endorotor | 16 month

CONTACTS AND LOCATIONS:
Overall Officials: frederic Prat, MD PHD, Principal Investigator — APHP
Locations (1):
- Hospital Beaujon, APHP, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided